CLINICAL TRIAL: NCT00019435
Title: Phase I Study of LMB-9, a Recombinant Disulfide Stabilized Immunotoxin for Advanced Carcinomas That Express Lewis Y Antigen
Brief Title: LMB-9 Immunotoxin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066180; NCI-98-C-0078A; NCI-MB-400; NCI-T98-0005; NCT00001691 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-05-06 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2007-04

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Lung Cancer; Pancreatic Cancer
Keywords: stage IV colon cancer; stage IV breast cancer; recurrent breast cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent non-small cell lung cancer; recurrent pancreatic cancer; recurrent colon cancer; stage IV esophageal cancer; recurrent esophageal cancer; recurrent bladder cancer; stage IV bladder cancer; stage IV non-small cell lung cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Biological: LMB-9 immunotoxin

SUMMARY:
RATIONALE: The LMB-9 immunotoxin may be able to locate tumor cells and kill them without harming normal cells. This may be an effective treatment for advanced solid tumors.

PURPOSE: Phase I trial to study the effectiveness of LMB-9 immunotoxin in treating patients who have advanced solid tumors that have not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effects and the pharmacokinetics of LMB-9 immunotoxin in patients with advanced solid tumors that express Lewis Y antigen. II. Evaluate the anti-tumor activity and the immunogenicity of this treatment regimen in these patients.

OUTLINE: This is a dose-escalation study. Patients receive LMB-9 immunotoxin IV over 30 minutes on days 1, 3, and 5. Patients with negative neutralizing antibody to LMB-9 immunotoxin with stable or responding disease receive additional courses every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of LMB-9 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional cohort of 6 patients may be treated at the MTD. Patients are followed at 1 month and then every 2 months thereafter.

PROJECTED ACCRUAL: Approximately 20-30 patients will be accrued within 12-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced solid tumor refractory to standard treatment or for which no effective standard therapy exists Bladder cancer Breast cancer Colon cancer Esophageal cancer Gastric cancer Non-small cell lung cancer Pancreatic cancer Evaluable or measurable disease B3 antigen present on more than 30% of tumor cells No prior or concurrent CNS metastasis Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: At least 3 months Hematopoietic: Granulocyte count greater than 1,200/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT less than 5 times upper limit of normal Albumin at least 3.0 g/dL No history of liver disease No positive hepatitis B or C antigen Renal: Creatinine no greater than 1.4 mg/dL Cardiovascular: No history of coronary artery disease No New York Association class II-IV heart disease No arrhythmia requiring treatment No contraindications to pressor therapy Pulmonary: FEV1 and FVC greater than 65% of predicted value Pulmonary function test required of patients with significant smoking history or possible pulmonary disease Other: No active peptic ulcer disease No known allergy to omeprazole No history of seizure disorders No other concurrent malignancy No concurrent medical or psychiatric condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosourea) and recovered Endocrine therapy: At least 3 weeks since prior hormonal therapy Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Ira Pastan, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States